CLINICAL TRIAL: NCT03182595
Title: Variability of Sulfotransferase 1A1 Activity in Humans: an Approach to Improve Predictive Drug Response - Part I: Analysis of Intraindividual Variation in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hospital da Luz, Portugal (Other)
Collaborators: Universidade Nova de Lisboa (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HLUZ_001_2016
Record Dates: First submitted 2017-05-25; First posted 2017-06-09 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- open---label (Experimental): An open---label, single centre, nonrandomized clinical study in healthy volunteers, with intervention over a 13---week period.
  Interventions: Drug: Paracetamol

INTERVENTIONS:
Drug: Paracetamol — Volunteers will be screened at visit 1, and if they meet the inclusion/exclusion criteria they will receive the intervention at visit 2. At visit 2, complying subjects will receive a tablet containing 1 gram of paracetamol and have a blood sample collected 2 hours after administration; these procedures will be repeated on 2 more occasions (visits 3 and 4). The subjects will come for 5 visits during the study. Visit 1 and 2 must occur within 7 days of each other, visits 2, 3 and 4 will be four weeks (± 3 days) apart and visit 5 scheduled four weeks (± 3 days) after visit 4.

SUMMARY:
An open-label, single centre, nonrandomized clinical study in healthy volunteers, with intervention over a 13---week period. After written informed consent, subjects will undergo screening evaluations (Visit 1). One week after visit 1, subjects who meet the selection criteria will enter a run---in period of 8 weeks where participants will receive paracetamol 1g tablet and collect a blood sample at monthly intervals (visits 2, 3 and 4). A final visit for safety assessment will take place at week 13 (visit 5). Blood samples will be used to quantify P, PG e PS.

DETAILED DESCRIPTION:
To be able to predict efficacy and adverse reactions involving compounds metabolized by sulfonation, the investigators need more information on SULTs. Studies of in vivo sulfonation in humans are lacking, although they are of key importance in assessing the functional consequences of individual variation. In our current study, the investigators will start by developing an HPLC method of quantifying SULT1A1 activity using paracetamol as probe substrate and studying intraindividual variation in healthy adults. Advantages of using paracetamol as a probe substrate for in vivo phenotyping of SULT1A1 include: wide safety margin for in vivo use, easy and ready administration of the drug, significant metabolism by the enzyme of interest, short half---life, linear pharmacokinetics over a wide concentration range and a limited number of metabolites, quantifiable in plasma.15,24 In a subsequent study, the investigators plan to study interindividual variation in a larger sample, including subjects with chronic disease and on medication.The investigators expect to provide a valuable new tool to explore the clinical significance of variation of SULT1A1 activity, the most important SULT on drug metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females, over 18 years of age,
* Informed of the nature of the study and giving written informed consent,
* Report no significant diseases during screening,
* Have normal CBC, renal function and liver enzymology,
* Have no contraindication for paracetamol,
* Be on no regular medical treatment, except for contraceptives,
* Be able to communicate effectively with study personnel.

Exclusion Criteria:

* Hypersensitivity or idiosyncratic reaction to paracetamol,
* Intake of any medication, except for contraceptives, within 14 days before start of the study,
* Pregnancy or breastfeeding,
* BMI <18 kg/m2,
* Participation in a clinical study of any investigational product 1 month prior to visit 1 or during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-03-17 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
- Coefficient of variation of paracetamol sulfonation index (PSI), a ratio between the measured plasma concentrations of paracetamol sulfate (PS) and PS+ paracetamol glucoronide (PG) + paracetamol (P) | 9 months

SECONDARY OUTCOMES:
Reproductibility, sensitivity and accuracy of the HPLC method (human samples will be used to validate the method); | 9 months
Relationships between PSI and subject characteristics (gender, age, genotype, smoking status, caffeine consumption, alcohol consumption, oral contraceptive use); | 9 months
Relationship between SULTA1 expression and predose and postdose metabolic profiles; | 9 months
Association between SULT1A1 genotype and SULT1A1 expression (optional); | 9 months
Association between PSI and SULT1A1 genotype (optional). | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Natália Marto, MD, Principal Investigator — Hospital da Luz
Locations (1):
- Hospital da Luz, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marto N, Morello J, Antunes AMM, Azeredo S, Monteiro EC, Pereira SA. A simple method to measure sulfonation in man using paracetamol as probe drug. Sci Rep. 2021 Apr 27;11(1):9036. doi: 10.1038/s41598-021-88393-3. PMID 33907224